CLINICAL TRIAL: NCT05250960
Title: Evaluating the Use of Pre-epidural Placement of Sequential Compression Devices (SCD) to Prevent Hypotension
Brief Title: Pre-epidural Sequential Compression Devices (SCDs) to Prevent Hypotension During Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 21-020
Record Dates: First submitted 2022-02-18; First posted 2022-02-22 (Actual); Results first posted 2025-03-03 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Hypotension; Labor Complication
MeSH Terms: conditions — Hypotension; Obstetric Labor Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Intervention - SCD arm (Experimental): Patient will receive 1L of LR and have SCDs applied 15 minutes before epidural placement and will be removed 1 hour after epidural placement
  Interventions: Device: SCD
- Control - no SCD arm (No Intervention): Patient will receive 1L of LR during and after epidural placement with no use of SCDs

INTERVENTIONS:
Device: SCD — Patient will receive 1L of LR and have SCDs applied 15 minutes before epidural placement and will be removed 1 hour after epidural placement
  Arms: Intervention - SCD arm

SUMMARY:
When hypotension is related to epidural placement, this can occur within 15-60 minutes after placement. The purpose of this study is to build upon this preliminary work and to use a randomized controlled trial to examine the effectiveness of SCDs in preventing hypotension among a larger sample of laboring women who receive an epidural analgesia. This study will use a randomized, non-blinded, controlled design with two arms:

* Arm 1: Patient will receive 1L of LR and have SCDs applied 15 minutes before epidural placement and will be removed 1 hour after epidural placement
* Arm 2: Patient will receive 1L of LR during and after epidural placement with no use of SCDs

DETAILED DESCRIPTION:
When hypotension is related to epidural placement, this can occur within 15-60 minutes after placement. The purpose of this study is to build upon this preliminary work and to use a randomized controlled trial to examine the effectiveness of SCDs in preventing hypotension among a larger sample of laboring women who receive an epidural analgesia. This study will use a randomized, non-blinded, controlled design with two arms:

* Arm 1: Patient will receive 1liter (L) of lactated ringers (LR) and have SCDs applied 15 minutes before epidural placement and will be removed 1 hour after epidural placement
* Arm 2: Patient will receive 1L of LR during and after epidural placement with no use of SCDs Outcome variables include occurrence of maternal hypotension or Category II fetal tracings in the first hour after epidural placement.

ELIGIBILITY:
Inclusion Criteria:

* Laboring at Bethesda North Hospital Labor & Delivery Unit
* Will receive epidural analgesia
* 37+ weeks gestation
* Singleton pregnancy
* Category 1 tracings only before epidural placement

Exclusion Criteria:

* Under 18 years old
* Does not speak English
* Unable to consent to involvement in the research study
* Diagnosed with fetal demise
* Diagnosis of pre-existing hypertension
* Diagnosis of gestational hypertension
* Diagnosis of pre-eclampsia
* Diagnosis of diabetes
* Breech presentation
* Contraindications to lower leg compression (ex: fractured bones in leg, cellulitis, lower limb amputation, etc.)
* Contraindications to receiving 1L of LR
* Blood pressure on admission systolic blood pressure (SBP)>160 or diastolic blood pressure (DBP)>110
* Fetal heart rate abnormalities before epidural

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Laboring women only
Enrollment: 109 (Actual)
Dates: Start 2021-09-16 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-02-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Bethesda North Hospital, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention - Sequential Compression Devices (SCD) Arm: Patient will receive 1liter (L) of Lactated Ringers (LR) and have SCDs applied 15 minutes before epidural placement and will be removed 1 hour after epidural placement
  SCD: Patient will receive 1L of LR and have SCDs applied 15 minutes before epidural placement and will be removed 1 hour after epidural placement
- Control - no Sequential Compression Devices (SCD) Arm: Patient will receive 1L of LR during and after epidural placement with no use of SCDs
Period: Overall Study
Arm/Group | Intervention - Sequential Compression Devices (SCD) Arm | Control - no Sequential Compression Devices (SCD) Arm
Started | 53 | 56
Completed | 53 | 56
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention - SCD Arm | Control - no SCD Arm | Total
Number analyzed (Participants) | 53 | 56 | 109
Age, Continuous [Mean (Full Range); unit: years] | 29.1 [19 to 43] | 28.5 [19 to 37] | 28.8 [19 to 43]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 56 | 109
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 53 | 56 | 109

OUTCOME MEASURES:

1. Primary Outcome: Hypotension
Description: SBP <90mmHg or an SBP decrease more than 20% from baseline (physiological measure obtained via sphygmomanometer)
Time Frame: 1 hour
Measure: Number; unit: participants
Arm/Group | Intervention - SCD Arm | Control - no SCD Arm
Number analyzed (Participants) | 53 | 56
participants | 4 | 4

2. Primary Outcome: Category II Tracings
Description: Category II fetal tracings - fetal heart tracings will be reviewed by two independent nurses who will document whether Category II tracings are present or not
  Category II tracings - The classification of Category II tracings includes the following:
  bradycardia with variability, tachycardia, minimal variability, no variability with no recurrent decelerations, marked variability, absence of induced accelerations even after fetal stimulation, recurrent variable decelerations with minimal or moderate baseline variability, prolonged decelerations lasting more than two minutes, but less than ten minutes, recurrent late decelerations with moderate variability, variable decelerations with other characteristics such as slow return to baseline, overshooting the baseline, or 'shoulders'
Time Frame: 1 hour
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention - SCD Arm | Control - no SCD Arm
Number analyzed (Participants) | 53 | 56
Participants | 17 | 13

ADVERSE EVENTS:
Time Frame: During delivery
Arm/Group | Intervention - SCD Arm | Control - no SCD Arm
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/56
Other Adverse Events (participants affected / at risk) | 0/53 | 0/56

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-27): https://cdn.clinicaltrials.gov/large-docs/60/NCT05250960/Prot_SAP_000.pdf